CLINICAL TRIAL: NCT06559397
Title: Proprioceptive Puzzle: The Effect of Cervical Proprioceptive Errors on Quantitative Sensory Tests and Body Awareness in Young Adults
Brief Title: Proprioceptive Puzzle: Effects on Quantitative Sensory Tests and Body Awareness
Status: Completed | Type: Observational
Sponsor: Nagihan Acet (Other)
Responsible Party: Sponsor-Investigator, Nagihan Acet, Asst. Prof., Atılım University
Organization: Atılım University (Other)
Other Study IDs: AtılımU-2
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cervical Proprioceptive Error in Healthy Young Individuals
Keywords: Cervical proprioception; Joint position sense; Pain; Temporal summation; Mechanosensitivity; Conditioned pain modulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proprioceptive deficit positive group: This group consists of young participants who exhibit a proprioceptive error in their cervical proprioception test. Proprioceptive error refers to an inaccurate perception of the head's position in space. In this study, participants with a deviation greater than 5 degrees during the test will be classified into this group.
  Interventions: Other: Assessment of cervical proprioception
- Proprioceptive deficit negative goup: This group includes young participants who do not show any proprioceptive error in the cervical proprioception test. These participants accurately perceive the position of their head and thus do not have a proprioceptive deficit (less than 5 degrees)
  Interventions: Other: Assessment of cervical proprioception

INTERVENTIONS:
Other: Assessment of cervical proprioception — Cervical proprioception will be assessed using the 'head position error test' in both right and left rotation directions with the CROM device. Participants will be then divided into two groups based on the presence of proprioceptive errors (>5°).

SUMMARY:
Background: Cervical proprioception, referring to the awareness of the head's position in space, plays a crucial role in maintaining postural control and preventing musculoskeletal injuries. While previous research has established the importance of cervical proprioception in motor function, its specific impact on body awareness and pain-related aspects remains less explored, particularly in healthy young individuals.

Aim: This prospective cross-sectional study aims to investigate the impact of cervical proprioceptive error on body awareness, pressure pain threshold, pressure pain tolerance, conditioned pain modulation, and temporal summation in healthy young individuals.

Methods: In asymptomatic participants, cervical proprioception will be assessed using the 'head position error test' in both right and left rotation directions with the CROM device. Participants will be then divided into two groups based on the presence of proprioceptive deviation (>5°). Body awareness will beassessed using the 'Body Awareness Questionnaire,' while pressure pain threshold, pain tolerance, and temporal summation will be measured bilaterally with an algometer device (2 cm lateral to the C2 and C7 spinal processes, midpoint of the upper part of the trapezius, and over the temporomandibular joint) in both groups. Subsequently, the two groups will be compared using independent samples t-tests.

DETAILED DESCRIPTION:
Cervical proprioception, which refers to the awareness of the head's position in space, is a fundamental component of postural control and the prevention of musculoskeletal injuries. This sense is mediated by sensory receptors located in the muscles, joints, and skin of the cervical spine, providing critical feedback for maintaining balance and coordinating movements. Previous studies have extensively documented the role of cervical proprioception in motor function, highlighting its importance in activities that require precise head and neck movements.

Despite these findings, there is a gap in the literature regarding the specific impact of cervical proprioception on body awareness and pain-related parameters in healthy individuals. Body awareness, or the conscious perception of body position and movement, is essential for efficient motor control and overall well-being. Additionally, understanding how proprioceptive errors in the cervical region might influence pain perception could provide insights into mechanisms underlying chronic pain conditions.

The primary aim of this prospective cross-sectional study is to investigate the impact of cervical proprioceptive error on body awareness, pressure pain threshold, pressure pain tolerance, conditioned pain modulation, and temporal summation in asymptomatic young individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-25 years old

Exclusion Criteria:

* History of cervical spine injuries or disorders
* Chronic pain conditions or diagnosed musculoskeletal disorders
* Previous neck or spine surgeries
* Neurological or psychiatric conditions affecting proprioception or pain perception
* Use of medications influencing pain sensitivity or proprioception
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study involves healthy young participants aged between 18 and 25 years. The participants will be divided into two groups based on the presence of cervical proprioceptive deviation (greater than 5°) as measured by the 'head position error test' using a CROM device.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Quantitative sensory testing | Immediately after the intervention
  Quantitative sensory testing including pain threshold, tolerance, conditioned pain modulation, and temporal summation will be assessed by pressure algometer. The "pain threshold" is the point at which a person first feels pain, the "pain tolerance" is the last point that a person can tolerate, and the "temporal summation" is the first painful threshold evaluated after 10 repeats of the pain threshold. Conditioned pain modulation is the modulation of pain perception under varying conditions. In the current study, a cold stimulus will be used.
Assessment of body awareness | Immediately after the intervention
  Body awareness will be assessed through a questionnaire, consisting of 18 items, divided into 4 subgroups aimed at determining the sensitivity level of normal or abnormal body composition (1. Changes during the body process, 2. Sleep-wake cycle, 3. Estimation of disease onset, 4. Prediction of bodily reactions). Participants are asked to rate each item on a scale of 1 to 7. The overall score is calculated, and a higher score indicates better body awareness. The validity and reliability of the questionnaire are reported to be high.

CONTACTS AND LOCATIONS:
Overall Officials: Nagihan Acet, Principal Investigator — Atılım University
Locations (1):
- Atılım University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044
- [Background] Kulkarni V, Chandy MJ, Babu KS. Quantitative study of muscle spindles in suboccipital muscles of human foetuses. Neurol India. 2001 Dec;49(4):355-9. PMID 11799407
- [Background] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Background] Mehling WE, Gopisetty V, Daubenmier J, Price CJ, Hecht FM, Stewart A. Body awareness: construct and self-report measures. PLoS One. 2009;4(5):e5614. doi: 10.1371/journal.pone.0005614. Epub 2009 May 19. PMID 19440300
- [Background] Yang J, Lee B, Kim C. Changes in proprioception and pain in patients with neck pain after upper thoracic manipulation. J Phys Ther Sci. 2015 Mar;27(3):795-8. doi: 10.1589/jpts.27.795. Epub 2015 Mar 31. PMID 25931733
- [Background] Law EY, Chiu TT. Measurement of cervical range of motion (CROM) by electronic CROM goniometer: a test of reliability and validity. J Back Musculoskelet Rehabil. 2013;26(2):141-8. doi: 10.3233/BMR-2012-00358. PMID 23640315
- [Background] Walton DM, Macdermid JC, Nielson W, Teasell RW, Chiasson M, Brown L. Reliability, standard error, and minimum detectable change of clinical pressure pain threshold testing in people with and without acute neck pain. J Orthop Sports Phys Ther. 2011 Sep;41(9):644-50. doi: 10.2519/jospt.2011.3666. Epub 2011 Sep 1. PMID 21885906
- [Background] Karaca, S. (2017). Vücut Farkındalığı Anketinin Türkçe uyarlaması: Geçerlik ve güvenirlik çalışması (Yayınlanmamış yüksek lisans tezi). Muğla Sıtkı Koçman Üniversitesi Sağlık Bilimleri Enstitüsü, Muğla.
- [Background] Heisler AC, Song J, Dunlop DD, Wohlfahrt A, Bingham CO III, Bolster MB, Clauw DJ, Marder W, Phillips K, Neogi T, Lee YC. Association of Pain Centralization and Patient-Reported Pain in Active Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2020 Aug;72(8):1122-1129. doi: 10.1002/acr.23994. Epub 2020 Jul 21. PMID 31162824
- [Derived] Acet N, Begen S. The proprioceptive puzzle: An observational study investigating the effects of cervical proprioceptive errors on quantitative sensory testing and body awareness in young individuals. PLoS One. 2025 Apr 21;20(4):e0321645. doi: 10.1371/journal.pone.0321645. eCollection 2025. PMID 40257972